CLINICAL TRIAL: NCT05330169
Title: Prospective Observational Cohort Study to Evaluate Hearing Toxicity Before and After Chemoradiotherapy in Patients With Nasopharyngeal Carcinoma
Brief Title: Hearing Impairment of Nasopharyngeal Carcinoma
Status: Completed | Type: Observational
Sponsor: Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Kai Hu, professor, Guangxi Medical University
Other Study IDs: GuangxiMUHK3
Record Dates: First submitted 2022-03-28; First posted 2022-04-15 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Hearing Toxicity; Chemoradiotherapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This observational cohort study was aimed to evaluate the hearing toxicity at multiple time points from baseline to 1 year after radical chemoradiotherapy among nasopharyngeal carcinoma patients.

DETAILED DESCRIPTION:
With the development of radiotherapeutic techniques and equipment as well as advances in treatment modalities, the 5-year overall survival of patients with non-disseminated NPC has exceeded 80%. However, the incidence of hearing toxicity did not decrease significantly compared with the past. The hearing loss remains the second most common toxicity after xerostomia. Audiometry, acoustic impedance testing, eustachian tube pressure measurements, and distortion product otoacoustic emissions will be used to compare hearing before treatment and up to 1 year after radical chemoradiotherapy. The related factors affecting the hearing of NPC patients will also be investigated and explored.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed non-keratinizing nasopharyngeal carcinoma(WHO II/III).
2. About to undergo radical chemoradiotherapy with intensity-modulated radiotherapy (IMRT).
3. Eastern Cooperative Oncology Group performance status≤1.
4. Adequate marrow function: neutrocyte count≥1.5×10e9/L, hemoglobin

   ≥90g/L, and platelet count≥100×10e9/L.
5. Alanine Aminotransferase (ALT)/Aspartate Aminotransferase (AST)

   ≤2.5×upper limit of normal (ULN), and bilirubin≤ 1.5×ULN.
6. Adequate renal function: creatinine clearance rate≥ 60 ml/min (Cockcroft-Gault formula).
7. Patients must be informed of the investigational nature of this study and give written informed consent.

Exclusion Criteria:

1. Age > 60 or < 18.
2. Receiving additional targeted therapy or immunotherapy except for radiotherapy and chemotherapy.
3. With a condition that could cause hearing impairment, such as ear canal cerumen blockage, ear canal foreign body blockage, cholesteatoma, tympanic membrane perforation, cholesteatoma otitis media, middle ear granulation tissue growth, inner ear labyrinthitis, sudden nerve deafness, Meniere's disease, acoustic neuroma, and so on.
4. Patients who received aminoglycoside antibiotics or macrocyclic lipid antibiotics (such as streptomycin, gentamicin, kanamycin, neomycin, tobramycin, minocycline, erythromycin, roxithromycin, etc.) orally or intravenously within 30 days before treatment.
5. Patients with hearing loss at the baseline（except for those with conductive hearing loss diagnosed by at least two deputy chief physicians as nasopharyngeal carcinoma-related）
6. Patients who received additional treatment during the observation period due to disease progression.
7. Pregnant or breastfeeding.
8. Patients with prior malignancy who have received systemic chemotherapy or head and neck radiotherapy.
9. Any other condition, including symptomatic heart failure, unstable angina, myocardial infarction, active infection requiring systemic therapy, mental illness or domestic/social factors, deemed by the investigator to be likely to interfere with a patient's ability to sign informed consent, cooperate and participate in the study, or interferes with the interpretation of the results.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: nasopharyngeal carcinoma patients
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Hearing level (decibel) | up to 16 months
  We will use pure tone audiometry to access the hearing level (decibel) before treatment and serially up to 1 year after radical chemoradiotherapy.
The ratio of distortion product otoacoustic emission(DPOAE) failure | up to 16 months
  We will use distortion product otoacoustic emission(DPOAE) to access the hearing before treatment and serially up to 1 year after radical chemoradiotherapy.

SECONDARY OUTCOMES:
The ratio of Eustachian tube dysfuction(ETD) | up to 16 months
  We will use eustachian tube pressure measurement to access the eustachian tube function before treatment and serially up to 1 year after radical chemoradiotherapy.
Tympanogram type | up to 16 months
  We will use acoustic impedance tests to access the tympanogram type before treatment and serially up to 1 year after radical chemoradiotherapy.

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi, China

IPD SHARING:
Plan to Share IPD: No